CLINICAL TRIAL: NCT04820790
Title: Mobile Application for Monitoring Patients With Home Oxygen. A Protocol of a Randomized and Controlled Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ToDoMed (Other)
Responsible Party: Principal Investigator, Anisbed Naranjo Rojas, Respiratory therapist - Magister, ToDoMed
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2021-03-20; First posted 2021-03-29 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Oxygen-therapy
Keywords: Oxygen-therapy; e-Health; Mobile applications
MeSH Terms: interventions — Amyloid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 1 (Experimental): The efficiency of the mobile app in the follow-up of patients with home oxygen will be evaluated during 3 months
  Interventions: Other: Mobile applications
- Intervention Group 2: (No Intervention): Regular monitoring of the home oxygen without mobile app during 3 months

INTERVENTIONS:
Other: Mobile applications — Monitoring of patients with home oxygen through a mobile application
  Other Names: App
  Arms: Experimental Group 1

SUMMARY:
The use of mobile technology has become part of the reality capable of changing the health services' paradigm. As a proof of that, nowadays, technology is seemed as a key tool in processes such as: data collection, epidemiological surveillance, health promotion, and disease prevention. Therefore, technological tools should be taken as an advantage to optimize the control or monitoring of patients with chronic diseases including those who require the use of home oxygen therapy.

Objective: Determine the efficiency of a mobile application for clinical monitoring of patients who require home oxygen therapy.

Methods A randomized-controlled clinical trial including individuals whose age is 18 years or older who have been diagnosed with Chronic Obstructive Pulmonary Disease (COPD) under treatment with home oxygen therapy. The sample will be divided in two groups: the intervention group will be made up of those who are followed up with the mobile app, and the control group will be made up of the patients who are followed up conventionally (regular visit of the respiratory caregiver). To measure the effect of the intervention, some outcomes variables will be taken as the recognition of self-management of dyspnea, number of exacerbations associated with oxygen therapy, and the frequency of underutilization of oxygen supplies.

DETAILED DESCRIPTION:
The Continuous Home Oxygen-therapy (abbreviated as OCD in Spanish) refers to the supply of oxygen for continuous, general, and/or indefinite use at the home of patients with chronic hypoxemia. The purpose of this treatment is to prolong the life of the hypoxemic patient, improve exercise tolerance, and control clinical deterioration due to low oxygen saturation.

Contextualizing the use of home oxygen in Colombia, it was observed that there was an increase in the prevalence of COPD (Chronic Obstructive Pulmonary Disease) as well as the prescription of home oxygen in the first phases of the treatment. It was found that 3.176 patients were enrolled in the home care program without knowing their sociodemographic and epidemiological characteristics. The reason behind is that there are few epidemiological studies that refer to this therapy. However, Gonzales M. et al. emphasize that current indications should be reviewed and research carried out in order to determine guidelines for recommending home oxygen in patients with COPD.

Methods / Design Study Design A randomized controlled clinical trial divided in two parallel groups with a 3-months duration will be performed in order to evaluate the efficiency of a mobile application used for the monitoring of patients with home oxygen. The control group will be made up of individuals with oxygen therapy undergoing regular monitoring (periodic visits by the respiratory caregiver), and the intervention group formed by those who have conventional monitoring with the use of the mobile app called AppO2.

Sample's size calculation A total of 32 individuals (16 for the experimental group and 16 for the control one) would be necessary to recruit, for a 1:1 ratio, a power of 80% (beta error = 20%), a certainty of 95% (alpha error = 5%) and assuming that the intervention in the experimental group will cause a 3% increase with a ±6 standard deviation in recognition of self-management of dyspnea. A final size of 44 individuals has been established (22 for the EG and 22 for the CG) to minimise the effect of possible losses in statistical power.

Intervention:

The control group comprises patients who will be under the conventional follow-up of clinical assessment and control of home oxygen supplies. The intervention group will be monitored conventionally, and they will additionally have a mobile app, "AppO2". We will follow a consecutive sampling. Patients will be recruit as on the go. The allocation will be randomly performed using a statistical software called EPIDAT, 3.1.

Study variables

The following results variables and independent variables are suggested to achieve the proposed objectives:

Variables:

* Oxygen saturation through a pulse oximeter, capillary filling, respiratory rate, heart rate, duration time of the oxygen cylinder.
* Oxygen saturation and inspired fraction of oxygen relationship
* Borg dyspnea scale
* Oxygen saturation and inspired fraction of oxygen relationship
* Recognition of self-management of dyspnea and quality of life through the mobile app.
* Saint George questionnaire for the assessment of health-related (CVRS) quality of life Statistical analysis A descriptive analysis of the variables under study will be carried out by characterising the patients. Also, graphs and frequency tables will be constructed for the qualitative variables, and the calculation of central tendency measures (mean), dispersion (standard deviation), and position (limits of the distribution and range) for the quantitative variables.

For the bivariate analysis, the Student's T-test will be performed to compare two means, while for the qualitative variables, the chi-square test and Fisher's exact test will be used. For the analysis of three or more means, the repeated measures analysis of variance (ANOVA) will be calculated. Multiple linear regressions will be used to adjust the App use's impact and eliminate confounding factors. The standardized beta coefficients, the adjusted coefficient of determination, the residuals, etc., will be calculated. An alpha error <5% will be accepted for all statistical analyses, and confidence intervals will be calculated for 95% confidence (95% CI). For the complete statistical analysis, SPSS Statistics software, version 25.0 (IBM Corp), will be used.

Practical applicability The general objective of this protocol is to evaluate the efficiency of a mobile application in the follow-up of patients with home oxygen therapy through an intervention aimed at reducing exacerbations. Besides, an attempt will be made to identify the adequacy of the prescription of oxygen systems and establish the underutilisation of oxygen supplies at home. A two-group randomized clinical follow-up will be used to evaluate the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of 18 years of age and older
* Patient with PaO2 <60 mmHg, SO2 <89% and dyspnea. Patients with home oxygen therapy enrolled in-home care programs during the study period.
* Time of evolution of the disease greater to one year
* Patients who express their willingness to participate in the study through their informed consent.

Exclusion Criteria:

Patients with the following exceptional situations will be excluded from the study:

* Patients with invasive and/or non-invasive mechanical ventilation
* Patients with the inability to operate a mobile application or those who do not have a smartphone with an operating system (Android or iOS) and available data connection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Recognition of self-management of dyspnea and through the mobile app. | up to 12 weeks
  The Borg scale is a visual analogue scale standardised and validated . It is quick and easy to apply, allowing a graphical evaluation of the subjective perception of respiratory distress by the same patient. It has been used since the 1970s and has a range from 0 to 10. The scale determines dyspnea intensity and has a written expression added to the number, which helps categorise dyspnea's sensation in the individual being tested. The result is recorded and encoded. The interval between the ranges of the scale increases progressively, and the number 10 shows the greatest perception of dyspnea. The maximum point indicates that the severity of the disease has increased even above 10.
Saint George questionnaire for the assessment of health-related quality of life | up to 6 weeks
  It consists of 50 items divided into three scales: symptoms, activity, and impact. The items on the symptom scale refer to the frequency and severity of respiratory symptoms. The items on the activity scale assess the limitation of the activities due to dyspnea. In the impact scale, the psychological and social functional disorders produced by the disease are assessed. The items are formulated in two different ways: in the form of a question with five multiple choices/answers in which just one can be selected, and in the form of a sentence with two options: yes/no. The questionnaire is preferably self-administered, although it is also accepted through a personal interview. The average completion time is 10 minutes. The score is calculated for each of the questionnaire scales, and there is also an overall score. The range of all is from 0 (without altering the quality of life) until 100 (maximum alteration of life quality).

OTHER OUTCOMES:
Oxygen saturation | up to 6 weeks
  Non-invasive measurement of oxygen carried by hemoglobin within blood vessels. It is performed with a device called a pulse oximeter, which continuously evaluates the oxygen saturation at the peripheral level. the oxygen pressure saturation shown by the device represents the average of the measurements obtained during the previous 3 to 6 seconds. Normal readings from a pulse oximeter should normally range from 95 to 100 percent. Values below 90 percent indicate hypoxemia and the need for supplemental oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Molina Recio, PhD, Study Director — Universidad de Córdoba - España; Luis A Pérula de torres, PhD, Study Director — Universidad de Córdoba - España
Locations (1):
- TodoMed, Palmira, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCoy RW. Options for home oxygen therapy equipment: storage and metering of oxygen in the home. Respir Care. 2013 Jan;58(1):65-85. doi: 10.4187/respcare.01932. PMID 23271820
- [Result] Bott J, Blumenthal S, Buxton M, Ellum S, Falconer C, Garrod R, Harvey A, Hughes T, Lincoln M, Mikelsons C, Potter C, Pryor J, Rimington L, Sinfield F, Thompson C, Vaughn P, White J; British Thoracic Society Physiotherapy Guideline Development Group. Guidelines for the physiotherapy management of the adult, medical, spontaneously breathing patient. Thorax. 2009 May;64 Suppl 1:i1-51. doi: 10.1136/thx.2008.110726. No abstract available. PMID 19406863
- [Result] Rabe KF, Watz H. Chronic obstructive pulmonary disease. Lancet. 2017 May 13;389(10082):1931-1940. doi: 10.1016/S0140-6736(17)31222-9. Epub 2017 May 11. PMID 28513453
- [Result] Branson RD. Oxygen Therapy in COPD. Respir Care. 2018 Jun;63(6):734-748. doi: 10.4187/respcare.06312. PMID 29794207
- [Result] Mesquita CB, Knaut C, Caram LMO, Ferrari R, Bazan SGZ, Godoy I, Tanni SE. Impact of adherence to long-term oxygen therapy on patients with COPD and exertional hypoxemia followed for one year. J Bras Pneumol. 2018 Sep-Oct;44(5):390-397. doi: 10.1590/S1806-37562017000000019. PMID 30517340
- [Result] Oh H, Rizo C, Enkin M, Jadad A. What is eHealth (3): a systematic review of published definitions. J Med Internet Res. 2005 Feb 24;7(1):e1. doi: 10.2196/jmir.7.1.e1. PMID 15829471
- [Result] Mirkovic J, Kaufman DR, Ruland CM. Supporting cancer patients in illness management: usability evaluation of a mobile app. JMIR Mhealth Uhealth. 2014 Aug 13;2(3):e33. doi: 10.2196/mhealth.3359. PMID 25119490
- [Result] Hallensleben C, van Luenen S, Rolink E, Ossebaard HC, Chavannes NH. eHealth for people with COPD in the Netherlands: a scoping review. Int J Chron Obstruct Pulmon Dis. 2019 Jul 26;14:1681-1690. doi: 10.2147/COPD.S207187. eCollection 2019. PMID 31440044
- [Result] Gurbeta L, Badnjevic A, Maksimovic M, Omanovic-Miklicanin E, Sejdic E. A telehealth system for automated diagnosis of asthma and chronical obstructive pulmonary disease. J Am Med Inform Assoc. 2018 Sep 1;25(9):1213-1217. doi: 10.1093/jamia/ocy055. PMID 29788482
- [Result] Rassouli F, Boutellier D, Duss J, Huber S, Brutsche MH. Digitalizing multidisciplinary pulmonary rehabilitation in COPD with a smartphone application: an international observational pilot study. Int J Chron Obstruct Pulmon Dis. 2018 Nov 23;13:3831-3836. doi: 10.2147/COPD.S182880. eCollection 2018. PMID 30538444
- [Result] Bitsaki M, Koutras C, Koutras G, Leymann F, Steimle F, Wagner S, Wieland M. ChronicOnline: Implementing a mHealth solution for monitoring and early alerting in chronic obstructive pulmonary disease. Health Informatics J. 2017 Sep;23(3):197-207. doi: 10.1177/1460458216641480. Epub 2016 Apr 21. PMID 27102885
- [Result] Nguyen HQ, Donesky-Cuenco D, Wolpin S, Reinke LF, Benditt JO, Paul SM, Carrieri-Kohlman V. Randomized controlled trial of an internet-based versus face-to-face dyspnea self-management program for patients with chronic obstructive pulmonary disease: pilot study. J Med Internet Res. 2008 Apr 16;10(2):e9. doi: 10.2196/jmir.990. PMID 18417444
- [Result] Hernandez-Reyes A, Camara-Martos F, Molina Recio G, Molina-Luque R, Romero-Saldana M, Moreno Rojas R. Push Notifications From a Mobile App to Improve the Body Composition of Overweight or Obese Women: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Feb 12;8(2):e13747. doi: 10.2196/13747. PMID 32049065
- [Result] Yang F, Wang Y, Yang C, Hu H, Xiong Z. Mobile health applications in self-management of patients with chronic obstructive pulmonary disease: a systematic review and meta-analysis of their efficacy. BMC Pulm Med. 2018 Sep 4;18(1):147. doi: 10.1186/s12890-018-0671-z. PMID 30180835
- [Result] Scott IA, Scuffham P, Gupta D, Harch TM, Borchi J, Richards B. Going digital: a narrative overview of the effects, quality and utility of mobile apps in chronic disease self-management. Aust Health Rev. 2020 Feb;44(1):62-82. doi: 10.1071/AH18064. PMID 30419185
- [Result] Early J, Gonzalez C, Gordon-Dseagu V, Robles-Calderon L. Use of Mobile Health (mHealth) Technologies and Interventions Among Community Health Workers Globally: A Scoping Review. Health Promot Pract. 2019 Nov;20(6):805-817. doi: 10.1177/1524839919855391. Epub 2019 Jun 10. PMID 31179777
- [Derived] Naranjo-Rojas A, Perula-de Torres LA, Cruz-Mosquera FE, Molina-Recio G. Efficacy and Acceptability of a Mobile App for Monitoring the Clinical Status of Patients With Chronic Obstructive Pulmonary Disease Receiving Home Oxygen Therapy: Randomized Controlled Trial. J Med Internet Res. 2025 Jan 6;27:e65888. doi: 10.2196/65888. PMID 39761550
- [Derived] Naranjo-Rojas A, Perula-de-Torres LA, Molina-Recio G. Patients, caregivers, and healthcare professionals' needs when designing the content of a mobile application for the clinical monitoring of patients with chronic obstructive pulmonary disease and home oxygen therapy: A user-centered design. Internet Interv. 2022 Jun 10;29:100552. doi: 10.1016/j.invent.2022.100552. eCollection 2022 Sep. PMID 35756891
- [Derived] Naranjo-Rojas A, Perula-de-Torres LA, Cruz-Mosquera FE, Molina-Recio G. Mobile application for monitoring patients under home oxygen therapy: a protocol for a randomized controlled trial. BMC Fam Pract. 2021 May 26;22(1):104. doi: 10.1186/s12875-021-01450-8. PMID 34039277